CLINICAL TRIAL: NCT05424458
Title: Changes of Dental Anxiety, Aesthetic Perception and Oral Health-related Quality of Life Related to Influencing Factors of Patients' Demographics After Anterior Implant Treatment
Brief Title: Effect of Anterior Implant Treatment on DA, Aesthetic Perception and OHRQoL Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Feilong Deng (Other)
Responsible Party: Sponsor-Investigator, Feilong Deng, Professor, Hospital of Stomatology, Sun Yat-Sen University
Organization: Hospital of Stomatology, Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: KQEC-2021-46-01
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Dental Anxiety; Aesthetic Perception; Oral Health-related Quality of Life
Keywords: dental anxiety; aesthetic perception; oral health-related quality of life; anterior implant treatment

STUDY DESIGN:
Intervention Model Description: The subjects completed the Modified Dental Anxiety Scale (MDAS), the Orofacial Esthetic Scale (OSE) and the Oral Health Impact Profile-14 (OHIP-14), before implant surgery and after definitive prosthesis placement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm (Experimental): Patients received routine examinations before surgery. The surgical procedures were performed by experienced experts. Immediate loading protocol was delivered if the insertion torque was over 35 N·cm; otherwise, removable restorations with submerged implants were applied. After a healing period of 3 to 6 months, a definitive screw-retained porcelain-fused-to-metal (PFM) or a CAD/CAM zirconia restoration were performed.
  In the first month after definitive prosthesis placement, patients were recalled to complete the MDAS, OES and OHIP questionnaires for the second time. Changes of overall MDAS, OSE and OHIP score were defined as the score after definitive prosthesis placement minus that before the treatment. Negative score changes indicated score decrease of the second questionnaire compared to the first one. Positive score changes indicated score increase.
  Interventions: Procedure: Anterior Implant Treatment

INTERVENTIONS:
Procedure: Anterior Implant Treatment — Patients received routine examinations before surgery. The surgical procedures were performed by experienced experts. Immediate loading protocol was delivered if the insertion torque was over 35 N·cm; otherwise, removable restorations with submerged implants were applied. After a healing period of 3 to 6 months, a definitive screw-retained porcelain-fused-to-metal (PFM) or a CAD/CAM zirconia restoration were performed.

SUMMARY:
Accumulating evidence has revealed the effects of anterior implant procedures on dental anxiety (DA), aesthetic perception and oral health-related quality of life (OHRQoL). However, few reported the changes and influencing factors of the above outcomes before and after anterior implant treatment. The aim of this study was to evaluate the changes of DA, aesthetic perception and OHRQoL related to influencing factors of patients' demographics after anterior implant treatment.

DETAILED DESCRIPTION:
The purpose of this prospective study was to evaluate the changes of DA, aesthetic perception and OHRQoL related to influencing factors of patients' age, gender and educational status after anterior implant treatment.

The subjects (n=39) included in this prospective study were recruited from those patients with anterior missing teeth at the Department of Oral Implantology, Guanghua School of Stomatology, Sun Yat-sen University.

Patients satisfying the following inclusion criteria were recruited: (1) age≥18 years old; (2) partially anterior edentulous jaws; (3) patients will be given an anterior implant surgery and implant-supported fixed rehabilitation; (4) patients could express themselves and communicate normally; (4) willing to participate in and accept investigation. Exclusion criteria were (1) use of anti-anxiety and painkillers within 1 year.; (2) mental and psychological diseases with poor emotional self-control; (3) a history of previous implant loss; (4) ongoing active infections by endodontic or periodontal problems of all the remaining teeth; (5) combined complex surgery including maxillary sinus augumentation, and large-block autogenous bone grafting.

Before implant surgery, all participants signed an informed consent form and were given sufficient time in the waiting room to answer the following three scales. The modified dental anxiety scale (MDAS) included five questions with a 5-category scale, ranging from 'not' to 'extremely'. The Orofacial Esthetics Scale (OES) is a scale that was designed by 8 items to evaluate the self-perception of aesthetic implant treatment (Ranged from 0 to 10 scores, 0 is 'Very dissatisfied' and 10 is 'Very satisfied'). The Oral Health Impact Profile (OHIP) is to measure OHRQoL, comprising 14 statements with 5 scores (1 = Not, 2 = Seldom, 3 = Sometimes, 4 = Often, 5 = Very often; total scores: 14-70). Influencing factors of patients' demographics including age, gender and educational status were obtained from the medical records.

Patients received routine examinations before surgery. The surgical procedures were performed by experienced experts. Immediate loading protocol was delivered if the insertion torque was over 35 N·cm; otherwise, removable restorations with submerged implants were applied. After a healing period of 3 to 6 months, a definitive screw-retained porcelain-fused-to-metal (PFM) or a CAD/CAM zirconia restoration were performed.

In the first month after definitive prosthesis placement, patients were recalled to complete the MDAS, OES and OHIP questionnaires for the second time. Changes of overall MDAS, OSE and OHIP score were defined as the score after definitive prosthesis placement minus that before the treatment. Negative score changes indicated score decrease of the second questionnaire compared to the first one. Positive score changes indicated score increase.

Data were collected and evaluated from the scales by two independent researchers. Data were calculated by descriptive statistics (mean, standard deviation) and were analyzed using the SPSS 25.0 software package (SPSS Inc., USA). Mann-Whitney U test was used to determine the score change before and after anterior implant treatment. Mann-Whitney U test (gender) and Kruskal-Wallis test by Bonferroni correction (age and educational status) were applied for the influencing factors evaluation based on the changes of overall MDAS, OSE and OHIP score. The level of significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years old
* partially anterior edentulous jaws
* patients will be given an anterior implant surgery and implant-supported fixed rehabilitation
* patients could express themselves and communicate normally
* willing to participate in and accept investigation

Exclusion Criteria:

* use of anti-anxiety and painkillers within 1 year
* mental and psychological diseases with poor emotional self-control
* a history of previous implant loss
* ongoing active infections by endodontic or periodontal problems of all the remaining teeth
* combined complex surgery including maxillary sinus augumentation, and large-block autogenous bone grafting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Changes of the modified dental anxiety scale (MDAS) before and after anterior implant treatment | Before implant surgery and in the first month after definitive prosthesis placement
  Dental anxiety levels changes between two time points. The modified dental anxiety scale (MDAS) included five questions with a 5-category scale, ranging from 'not' to 'extremely'. On MDAS questionnaire numbers correspond to the dimensions (1 = Not, 2 = Slightly, 3 = Fairly, 4 = Very, 5 = Extremely. Overall MDAS score: Q1-Q5 summary score.).
Changes of the Orofacial Esthetics Scale (OES) before and after anterior implant treatment | Before implant surgery and in the first month after definitive prosthesis placement
  Aesthetic perception changes changes between two time points. The Orofacial Esthetics Scale (OES) is a scale that was designed by 8 items to evaluate the self-perception of aesthetic implant treatment (Ranged from 0 to 10 scores, 0 is 'Very dissatisfied' and 10 is 'Very satisfied').
Changes of the Oral Health Impact Profile (OHIP) before and after anterior implant treatment | Before implant surgery and in the first month after definitive prosthesis placement
  Oral health-related quality of life changes between two time points. The Oral Health Impact Profile (OHIP) is to measure OHRQoL, comprising 14 statements with 5 scores (1 = Not, 2 = Seldom, 3 = Sometimes, 4 = Often, 5 = Very often; total scores: 14-70).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Stomatology, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data may be available once published within one year.
Access Criteria: Sun Yat sen University RDD platform once the data are published.

REFERENCES:
- [Background] Kan JYK, Rungcharassaeng K, Deflorian M, Weinstein T, Wang HL, Testori T. Immediate implant placement and provisionalization of maxillary anterior single implants. Periodontol 2000. 2018 Jun;77(1):197-212. doi: 10.1111/prd.12212. Epub 2018 Feb 25. PMID 29478284
- [Background] Wang Y, Baumer D, Ozga AK, Korner G, Baumer A. Patient satisfaction and oral health-related quality of life 10 years after implant placement. BMC Oral Health. 2021 Jan 14;21(1):30. doi: 10.1186/s12903-020-01381-3. PMID 33446161
- [Background] Zhang X, Wang B, Qiao SC, Gu YX, Shi JY, Lai HC. A study on the prevalence of dental anxiety, pain perception, and their interrelationship in Chinese patients with oral implant surgery. Clin Implant Dent Relat Res. 2019 Jun;21(3):428-435. doi: 10.1111/cid.12779. Epub 2019 Apr 26. PMID 31025495
- [Background] Yoshida T, Masaki C, Komai H, Misumi S, Mukaibo T, Kondo Y, Nakamoto T, Hosokawa R. Changes in oral health-related quality of life during implant treatment in partially edentulous patients: A prospective study. J Prosthodont Res. 2016 Oct;60(4):258-264. doi: 10.1016/j.jpor.2016.01.010. Epub 2016 Mar 8. PMID 26968266
- [Background] Persic S, Celebic A. Influence of different prosthodontic rehabilitation options on oral health-related quality of life, orofacial esthetics and chewing function based on patient-reported outcomes. Qual Life Res. 2015 Apr;24(4):919-26. doi: 10.1007/s11136-014-0817-2. Epub 2014 Oct 8. PMID 25294397
- [Background] Bovaira M, Herrero Babiloni A, Jovani M, Penarrocha-Diago M, Gonzalez-Lemonnier S, Penarrocha-Oltra D. Preoperative Anxiety and Its Influence on Patient and Surgeon Satisfaction in Patients Receiving Dental Implant Surgeries Performed Under Intravenous Conscious Sedation. Int J Oral Maxillofac Implants. 2017 Jul/Aug;32(4):912-918. doi: 10.11607/jomi.5712. PMID 28708923
- [Background] Elfadil S, Johnston B, Normand C, Allen F, O'Connell B. An Investigation of the Characteristics of Edentulous Patients Who Choose or Refuse Implant Treatment. Int J Prosthodont. 2021 March/April;34(2):147-153. doi: 10.11607/ijp.6222. Epub 2020 Jun 26. PMID 32589000
- [Background] Sanchez-Perez A, Nicolas-Silvente AI, Sanchez-Matas C, Molina-Garcia S, Navarro-Cuellar C, Romanos GE. Primary stability and PES/WES evaluation for immediate implants in the aesthetic zone: a pilot clinical double-blind randomized study. Sci Rep. 2021 Oct 8;11(1):20024. doi: 10.1038/s41598-021-99218-8. PMID 34625591
- [Background] Bersezio C, Martin J, Herrera A, Loguercio A, Fernandez E. The effects of at-home whitening on patients' oral health, psychology, and aesthetic perception. BMC Oral Health. 2018 Dec 11;18(1):208. doi: 10.1186/s12903-018-0668-2. PMID 30537968
- [Background] Nielsen HB, Schou S, Bruun NH, Starch-Jensen T. Professional and patient-reported outcomes of two surgical approaches for implant-supported single-crown restoration: 1-year results of a randomized controlled clinical trial. Clin Oral Implants Res. 2022 Feb;33(2):197-208. doi: 10.1111/clr.13883. Epub 2021 Dec 17. PMID 34866250
- [Derived] Xie X, Zhang Z, Zhou J, Deng F. Changes of dental anxiety, aesthetic perception and oral health-related quality of life related to influencing factors of patients' demographics after anterior implant treatment: a prospective study. Int J Implant Dent. 2023 Aug 2;9(1):22. doi: 10.1186/s40729-023-00486-y. PMID 37530855